CLINICAL TRIAL: NCT05403138
Title: A Multi-center, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of Daratumumab in Patients With Anti-Aquaporin 4 Antibody Positive Neuromyelitis Optica Spectrum Disorders (NMOSD)
Brief Title: Safety and Efficacy of Daratumumab in Patients With Anti-Aquaporin 4 Antibody Positive Neuromyelitis Optica Spectrum Disorders
Acronym: DAWN
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022023
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder; NMO Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — daratumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daratumumab (Experimental): Induction Period: Participants received daratumumab (8mg/kg) via intravenous (IV) every 2 weeks for two cycles. This was followed by the Maintenance Period: Participants received daratumumab (4mg/kg) via IV infusion every 4 weeks from the third dose (Week 4) onwards.
  Interventions: Drug: Daratumumab
- Placebo (Placebo Comparator): Placebo contains the same buffer components without the active ingredient. Induction Period: Participants received matching placebo (8mg/kg) via intravenous (IV) every 2 weeks for two cycles. This was followed by the Maintenance Period: Participants received matching placebo (4mg/kg) via IV infusion every 4 weeks from the third dose (Week 4) onwards.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daratumumab — Induction Phase: (8mg/kg) via intravenous (IV) evey 2 weeks for two cycles. Maintenance Phase: (4mg/kg) IV every 4 weeks.
  Other Names: Darzalex
  Arms: Daratumumab
Drug: Placebo — Induction Phase: matching placebo (8mg/kg) via intravenous (IV) every 2 weeks for two cycles; Maintenance Phase: matching placebo (4mg/kg) IV every 4 weeks.
  Arms: Placebo

SUMMARY:
The objectives of this time-to-event study are to assess the efficacy and safety of Daratumumab as compared with placebo in participants with neuromyelitis optica spectrum disorder (NMOSD) who are anti-aquaporin-4 (AQP4) antibody-positive. NMOSD is an autoimmune disease of the central nervous system that predominantly affects the spinal cord, optic nerves, and area postrema. It is usually mediated by the pathogenic AQP4-IgG. Antibody-secreting cells (ASCs) have been recognized as essential sources of AQP4-IgG. CD38 is a glycoprotein that is highly expressed on ASCs. Daratumumab, a CD38-directed monoclonal antibody, has been shown to decrease the levels of autoantibodies in lupus, myasthenia gravis, or autoimmune encephalitis. This randomized controlled study aims to evaluate the therapeutic potential of daratumumab in NMOSD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥ 18 years old.
2. Diagnosis of NMO or NMOSD.
3. Anti-AQP4 antibody seropositive.
4. Historical relapse of at least 1 relapses in the last 12 months or 2 relapses in the last 24 months with at least 1 relapse in the 12 months prior to the screening.
5. Expanded Disability Status Scale score ≤ 7.5.
6. Patients must give written informed consent.

Exclusion Criteria:

1. Use of intravenous steroid pulse therapy or intravenous immunoglobulin or plasma exchange/adsorption within 3 weeks prior to Screening.
2. Use of tocilizumab, satralizumab, belimumab, ofatumumab within 1 months prior to Screening.
3. Patients treated with oral immunosuppressive agents other than steroids (e.g. azathioprine, mycophenolate mofetil, methotrexate, tacrolimus, cyclosporine in the 3 months prior to allocation.
4. Use of rituximab or inebilizumab within 6 months prior to Screening.
5. Patients infected with hepatitis B or C virus, or human immunodeficiency virus, or those having active infectious diseases.
6. Patients with a severe chronic infection or a history of recurrent infections.
7. Patients with a history of radiation treatment (whole body irradiation or lymphoid irradiation) or stem cell transplantation.
8. Patients who are pregnant or breast-feeding.
9. Patients who are participating in other clinical trials for NMOSD.
10. Patients diagnosed with cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Participants With An Adjudicated On-trial Relapse | Baseline, Up To 52 Weeks (End of Study)
  An On-trial Relapse was defined as a new onset of neurologic symptoms or worsening of existing neurologic symptoms with an objective change (clinical sign) on neurologic examination that persisted for more than 24 hours as confirmed by the treating physician. An adjudicated On-trial Relapse was defined by the protocol and positively adjudicated by the relapse adjudication committee.

SECONDARY OUTCOMES:
Adjudicated On-trial Annualized Relapse Rate (ARR) | Baseline, Up To 52 Weeks (End of Study)
  The adjudicated On-trial ARR was computed as the total number of relapses divided by the total number of patient years in the study period. A central independent committee was used to adjudicate all On-trial Relapses as determined by the treating physician. Results reported as adjusted adjudicated On-trial ARR based on a Poisson regression adjusted for randomization strata and historical ARR in 24 months prior to Screening.
Percentage of Participants With Worsening in Expanded Disability Severity Scale (EDSS) Score From Baseline to the end of study | Baseline, Up To 52 Weeks (End of Study)
  Disease-related disability was measured by the EDSS. The EDSS was an ordinal clinical rating scale that ranges from 0 (normal neurologic examination) to 10 (death) in half-point increments. A decrease in score indicates improvement.
Change From Baseline in Best Corrected Binocular Visual Acuity to the end of study | Baseline, Up To 52 Weeks (End of Study)
  Best corrected binocular visual acuity was measure with Early Treatment Diabetic Retinopathy Study (ETDRS) chart held at a distance of 2.52 meters.
Change From Baseline in Low-Contrast Visual Acuity Binocular Score to the end of study | Baseline, Up To 52 Weeks (End of Study)
  Low-contrast visual acuity test was used to determine the number of letters that can be read on a standardized low-contrast retro-illuminated 2.5% Sloan letter chart held at a distance of 2.52 meters. Binocular score was the number of letters read correctly on the chart using both eyes simultaneously. The total score ranges from 0-70. Higher score indicates better vision.
Blood AQP4-IgG Concentration Over Time | Baseline, Weeks 2, 4, 8, 12, 24, 48
  Blood AQP4-IgG Concentration was measured by Cell-Based Assay (CBA).
Percentage of Blood Antibody-Secreting Cells (ASCs) Over Time | Baseline, Weeks 2, 4, 8, 12, 24, 48
  Percentage of Blood ASCs was measured by flow cytometry.
Percentage of Blood Neurofilament Light Chain (NFL) Over Time | Baseline, Weeks 2, 4, 8, 12, 24, 48
  Percentage of Blood NFL was measured with Simoa (Single-molecule array).
Percentage of Blood Glial Fibrillary Acidic Protein (GFAP) Over Time | Baseline, Weeks 2, 4, 8, 12, 24, 48
  Percentage of Blood GFAP was measured with Simoa (Single-molecule array).
Change From Baseline In Modified Rankin Scale (mRS) Score At End Of Study | Baseline, Up To 52 Weeks (End of Study)
  Disease-related disability was measured by the mRS score. The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered from a neurological disability. The scale ranges from 0 (no disability) to 6 (death) in whole-point increments. A decrease in score indicates improvement.
Change From Baseline In Hauser Ambulation Index (HAI) Score At End of Study | Baseline, Up To 52 Weeks (End of Study)
  The HAI was used to evaluate gait and assess the time and effort used by the participant to walk 25 feet (8 meters). The scale ranges from 0 to 9, with 0 being the best score (asymptomatic; fully ambulatory with no assistance) and 9 being the worst (restricted to wheel chair; unable to transfer self independently). A decrease in score indicates improvement.
Change From Baseline In European Quality Of Life (EuroQoL) Health 5-Dimension Questionnaire (EQ-5D) Visual Analogue Scale At End Of Study | Baseline, Up To 52 Weeks (End of Study)
  The EuroQoL EQ-5D was a generic, standardized, self-administered instrument that provides a simple, descriptive profile and a single index value for health status. Assessments were made using the EQ-5D Visual Analogue Scale, which captures the self-rating of current health status using a visual "thermometer" with the endpoints of 100 (best imaginable health state) at the top and zero (worst imaginable health state) at the bottom. An increase in score indicates improvement.
Change From Baseline In EuroQoL EQ-5D Index Score At End Of Study | Baseline, Up To 52 Weeks (End of Study)
  The EuroQoL EQ-5D was a generic, standardized, self-administered instrument that provides a simple, descriptive profile and a single index value for health status. Index scores range from less than 0 to 1, with higher scores representing a better health status.
Change From Baseline in Speed of Timed 25-Foot Walk (T25W) at 24 Week Intervals During the DB Period | Baseline, Up To 52 Weeks (End of Study)
  The T25W was an assessment of walking ability. The time (in seconds) that the participant took to walk 25 feet was measured. Speed is calculated as 1/Timed 25-Foot Walk where time is measured in seconds. A positive change from baseline indicates an improvement.
Number of Participants With Adverse Events (AEs) | Baseline, Up To 52 Weeks (End of Study)
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Number of Participants With Adverse Events Serious Adverse Events (SAEs) | Baseline, Up To 52 Weeks (End of Study)
  A SAE was any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No